CLINICAL TRIAL: NCT05451121
Title: Comparing Effect of Propofol, Dexmedetomidine and Their Combination on Duration Mechanical Ventilation in Patient After Cardiac Surgery
Brief Title: Effect of Sedation Strategy on Duration Mechanical Ventilation in Patient After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anesthesia Research Group UA (Other)
Responsible Party: Principal Investigator, Plechysta Yelyzaveta, Chief of the anesthesia department, Anesthesia Research Group UA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0120U100656
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Failure; Mechanical Ventilation Complication; Sedation Complication
Keywords: LOHS, sedation, cardiac surgery, intensive care unit
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propofol (Experimental): Patient sedation after cardiac surgery at the intensive care unit. Continuous infusion of propofol (hypnotic agent) using a syringe pump at the dose of 1-1.5 mg / kg / h
  Interventions: Drug: Propofol
- Dexmedetomidine (Experimental): Patient sedation after cardiac surgery at the intensive care unit. continuous infusion of Dexmedetomidine (selective α2-adrenergic receptor (α2-AR) agonist) using a syringe pump at the dose of 0.5-1.0 mcg/ kg / h
  Interventions: Drug: Dexmedetomidine
- propofol and dexmedetomidine (Experimental): Patient sedation after cardiac surgery at the intensive care unit. Continuous infusion of propofol using a syringe pump at the dose of 0.5-1.5 mg / kg / h and dexmedetomidine 0.2-0.7 mcg\kg\h
  Interventions: Drug: Propofol and dexmedetomidine

INTERVENTIONS:
Drug: Propofol — patient sedation with a propofol (sedative agent) after cardiac surgery
  Arms: propofol
Drug: Dexmedetomidine — patient sedation with dexmedetomidine (selective α2-adrenergic receptor (α2-AR) agonist) after cardiac surgery
  Arms: Dexmedetomidine
Drug: Propofol and dexmedetomidine — Patients sedation with a drug combination: propofol and dexmedetomidine (selective α2-adrenergic receptor (α2-AR) agonist)
  Arms: propofol and dexmedetomidine

SUMMARY:
There is a direct relationship between the sedative agent and the duration of ventilation.

DETAILED DESCRIPTION:
Sedation and sedative agent have direct correlation to the mechanical length. As known mechanical length could increase length of the hospital stay (LOHS) and mortality rate. The right sedative agent can decrease the length go the mechanical ventilation. The goal of the research to compare 3 sedation strategies and their influence to the duration of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Multi vascular lesions of the coronary arteries according to coronary angiography;
* Heart valve damage was confirmed by, which is subject to surgical correction (aortic stenosis of III degree with a gradient on the aortic valve of more than 42 mmHg, aortic insufficiency III, mitral valve stenosis II-III, mitral regurgitation II-III)
* Age of patients from 18-80 years; • Patient consent to participate in the study;

Exclusion Criteria:

* Refusal to participate;

  * Hypersensitivity to propofol, dexmedetomidine;
  * Prolonged mechanical ventilation in case of surgical complications (bleeding, inadequate perfusion of the myocardium);
  * Occurred ischemic stroke;
  * History of the ischemic stroke;
  * History of the neurodegenerative diseases;
  * History of the mental disorders;
  * Use of neuroleptics, antidepressants for the last 5 years;
  * History of the cardiac surgery in the past;
  * Patients with chronic pulmonary disease (GOLD 3-4)
  * Patients with asthma (moderate or severe),
  * Participation in any other clinical trial;
  * Chronic renal failure (ClCr less than 50 ml / h)
  * Acute renal failure that occurred during surgery (ClCr less than 50 ml / h, or a decrease in the rate of diuresis to 0.1 ml / h in the first 4 hours after surgery and does not respond to diuretic therapy)
  * Chronic hepatic insufficiency if there are laboratory signs of hypo coagulation without the use of anticoagulant therapy (INR> 1.5)
  * If the patient has not stopped taking anticoagulants or antiplatelet agents in the preoperative period: warfarin 5 days before surgery, clopidogrel 5-7 days before surgery, xarelto / pradaxa 3 days before surgery),
  * History of the hematological disease;
  * Alcohol abuse in the anamnesis (3-4 times a week).
  * Condition after chemotherapy;
  * Pregnancy, lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
length of the mechanical ventilation | after cardiac surgery till extubation (up to first 24 hour after surgery)
  measure the length of the mechanical ventilation

SECONDARY OUTCOMES:
Length of the ICU stay | at the day of discharge of ICU (assessed up to day 5)
  thе amount of the days spent in the ICU
Length of the hospital stay | at the day of discharge of hospital (assessed up to day 5)
  thе amount of the days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yelyzaveta Plechysta, Study Chair — Chief of the anesthesia department
Locations (1):
- Anesthesia department Medical Network Dobrobut, Kyiv, Ukraine